CLINICAL TRIAL: NCT06845709
Title: Effects of Otago Exercises and Gaze Stabilization Exercises on Balance, Gait and Quality of Life in Elderly Stroke Patients
Brief Title: Effects of Otago and Gaze Stabilization Exercises on Balance, Gait and QOL in Elderly Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0237
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Balance; Distorted; Gait, Hemiplegic; Quality of Life
Keywords: Balance; Distorted; Gait, Hemiplegic; Quality of Life
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Patients will be divided in group A will receive Gaze Stabilization Exercises with conventional baseline treatment and group B patients will receive Otago Exercises with conventional baseline treatment. Patients will receive treatment of 40 minutes per session for 5 days a week for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gaze stabilization exercise (Experimental): Patients in group A will receive Gaze Stabilization Exercises with conventional baseline treatment
  Interventions: Other: gaze stabilization exercise
- otago exercise (Active Comparator): Patients in group B will receive Otago Exercises with conventional baseline treatment.
  Interventions: Other: otago exercise

INTERVENTIONS:
Other: gaze stabilization exercise — Patients in group A will receive Gaze Stabilization Exercises with conventional baseline treatment
  Arms: gaze stabilization exercise
Other: otago exercise — group B patients will receive Otago Exercises with conventional baseline treatment
  Arms: otago exercise

SUMMARY:
To compare effects of otago exercises and Gaze stabilization exercises on Balance, gait and quality of Life in elderly stroke patients

DETAILED DESCRIPTION:
Study design will be a randomized clinical trial . Total 46 stroke patients will be recruited from Riphah Rehabilitation center and General hospital, Lahore by using non-probability convenience sampling technique. Patients will be randomized and allocated into two intervention groups based on inclusion and exclusion criteria. Patients in group A will receive Gaze Stabilization Exercises with conventional baseline treatment and group B patients will receive Otago Exercises with conventional baseline treatment. Patients will receive treatment of 40 minutes per session for 5 days a week for 8 weeks. Berg Balance Scale, Dynamic Gait Index and Stroke specific quality of life will be used as assessment tools. Data will be analyzed by using SPSS 26 version.

ELIGIBILITY:
Inclusion Criteria:

* Had ischemic or haemorrhagic stroke ≤6 months
* Berg Balance Scale (BBS) score between 35 and 45
* Dynamic Gait Index score between 11 and 19
* Mini-mental status exam scores > 24

Exclusion Criteria:

* Participants with severe vision or hearing impairment
* Neurological disorders including epilepsy, Alzheimer's disease, vertigo, Parkinson disease, and stroke, muscular disorders which limit functional activity (OA, RA, etc)
* Medications that affect balance, severe cardiovascular conditions, recent lower limb injury or surgery
* Peripheral vestibular disorder

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | 10 months
  Berg Balance Scale Most reliable balance measuring tools for people suffered from stroke known as Berg Balance Scale. There are 14 questions in it, which aims at testing balance while sitting, standing, or performing specific movements. The total score on the Berg Balance Scale ranges from 0 to 56. 41-56: Have good balance and are at a low risk of falling. 21-40: Individuals have an increased risk of falling and may benefit from interventions to improve balance. 0-20: Individuals in this range have a significant balance impairment and are at a high risk of falling, requiring more intensive intervention and possibly assistance with mobility. Most of researches supported the validity and reliability of the BBS especially with stroke patients with high interclass correlation coefficients (ICCs) 0. 90
Dynamic Gait Index | 10 months
  Dynamic Gait Index A tool for assessing gait, balance and fall risk in stroke patients is known as Dynamic Gait Index. It involves eight generic movements that are representative of common gait problems like turning the head while walking, stepping over an object, or changing speed. Consist of total 0-24 score . Between 22-24: Normal and < 19: Abnormal. Scores below 19 are indicative of gait dysfunction . Dynamic Gait Index validity is 0. 90. The overall reliability was high (overall intra-class correlation coefficient = .96
Stroke-Specific Quality of Life (SS-QOL) | 10 months
  Stroke-Specific Quality of Life (SS-QOL) is a specially developed tool for estimating the quality of life of stroke survivors. SS-QOL scale consists of 49 items, comprises 12 domains include Energy, Family Roles, Language, Mobility, Mood, Personality, Self-care, Social Roles, Thinking, Upper Extremity Function, Vision, and Work/Productivity. Each item is scored on a 5-point Likert scale. where 1 indicates the most severe impairment and 5 indicates no impairment. The total score can range from 49 to 245, with higher scores representing better quality of life. In the SS-QOL domains, the Cronbach's alpha coefficients are generally provided with values of between 0. 73 and 0. 96. Concurrent validity was high with r = 0.94-0.95

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Vincenzo O, Luisi MLE, Alicante P, Ballarin G, Biffi B, Gheri CF, Scalfi L. The Assessment of the Risk of Malnutrition (Undernutrition) in Stroke Patients. Nutrients. 2023 Jan 29;15(3):683. doi: 10.3390/nu15030683. PMID 36771390
- [Background] Mead GE, Sposato LA, Sampaio Silva G, Yperzeele L, Wu S, Kutlubaev M, Cheyne J, Wahab K, Urrutia VC, Sharma VK, Sylaja PN, Hill K, Steiner T, Liebeskind DS, Rabinstein AA. A systematic review and synthesis of global stroke guidelines on behalf of the World Stroke Organization. Int J Stroke. 2023 Jun;18(5):499-531. doi: 10.1177/17474930231156753. Epub 2023 Mar 1. PMID 36725717
- [Background] Sim J, Shin C. Two stroke education programs designed for older adults. Geriatr Nurs. 2024 Jan-Feb;55:105-111. doi: 10.1016/j.gerinurse.2023.10.014. Epub 2023 Nov 17. PMID 37979469